CLINICAL TRIAL: NCT05230303
Title: Acute Effects of Caffeine Supplementation on Resistance Training Volume and Blood Antioxidant Status in Resitance Trained Men
Brief Title: Caffeine Supplementation, Resistance Training and Blood Antioxidant Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other)
Responsible Party: Principal Investigator, Aleksandra Filip-Stachnik, PhD, The Jerzy Kukuczka Academy of Physical Education in Katowice
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 01_2021
Record Dates: First submitted 2022-01-14; First posted 2022-02-08 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Caffeine
Keywords: sports performance, resistance training, nutrition, athlete

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine supplementation (Experimental): Group taking 3 mg/kg of caffeine
  Interventions: Dietary Supplement: Caffeine supplementation
- Placebo treatment (Placebo Comparator): Group taking placebo
  Interventions: Dietary Supplement: Placebo treatment

INTERVENTIONS:
Dietary Supplement: Caffeine supplementation — Two identical experimental sessions with a one-week interval between sessions (to allow complete recovery and ensure substance wash-out) will be taken. During the experimental sessions, participants will ingest caffeine in dose of 3 mg/kg of body mass. Caffeine will be provided in capsules containing the individual amount of caffeine and will be administered orally 60 min before the onset of the exercise protocol.
  Arms: Caffeine supplementation
Dietary Supplement: Placebo treatment — The experimental procedure for each particpant will include placebo supplementation. The manufacturer of the caffeine capsules will also prepare identical placebo capsules filled out with a microcrystalline cellulose. Placebo will be administered orally 60 min before the onset of the exercise protocol.
  Arms: Placebo treatment

SUMMARY:
The purpose of this study is to verify the effect of acute caffeine intake on resistance training volume and blood antioxidant status, in a randomised, double-blind, placebo-controlled crossover trial.

DETAILED DESCRIPTION:
Caffeine is one of the most commonly consumed psychoactive substances in the world. Several previous studies confirmed that caffeine improves several aspects of exercise performance, including resistance training outcomes. Interestingly, caffeine and its catabolic products, theobromine and xanthine, exhibit antioxidant and prooxidant properties. Additionally, resistance training promotes the generation of reactive oxygen species, which are important for the cellular adaptation process.

Hovewer, to the best of our knowledge, there is no information as to how caffeine combined with resistance training affects blood antioxidant status. Therefore, the aim of this study was to examine acute effects of caffeine supplementation on resistance training volume and blood antioxidant status in resistance trained men.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate,
* medical permission by physician
* "resistance-trained," defined as having a minimum of two years of resistance training experience
* minimum of 2 workout sessions per week in the last 6 months

Exclusion Criteria:

* neuromuscular or musculoskeletal disorders
* current injury
* using any medications, dietary supplements or ergogenic aids which could potentially affect the study outcomes
* a positive smoking status
* potential allergy to caffeine

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change the levels of oxidative stress markers | Day 1, Day 2
  Serum will be obtained for TOS/TOC (total oxidative stress), MDA (malondialdehyde), oncentration of TAS (total antioxidant status), activity of superoxide dismutase (SOD), catalase (CAT), glutathione peroxidase (GPx); concentartion of GSH (reduced glutathione) and UA (uric acid)
Changes in markers of muscle damage | Day 1, Day 2
  Serum will be obtained for activity of creatine kinase (CK) and lactate dehydrogenase (LDH), concentration of myoglobin (Mb)
Changes in Inflammation markers | Day 1, Day 2
  Serum will be obtained for level of interleukin 6, TNF alfa (tumor matrix factor), CRP (C-reactive protein)
Changes in markers of liver function | Day 1, Day 2
  Serum will be obtained for activity of ASPAT (aspartate aminotransferase), ALAT (alanine aminotransferase) and gamma glutamyltransferase (GGT)

SECONDARY OUTCOMES:
Changes in resistance training volume | During caffeine and placebo treatment
Changes in rate of perceived exertion after resistance training | Immediately after exercise protocol during caffeine and placebo treatment
Changes in heart rate during resistance training | During caffeine and placebo treatment
Changes in muscle soreness | prior to exercise, and 24, 48, 72, 96 and 120 hours post exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Zając, Profesor, Study Director — The Jerzy Kukuczka Academy of Physical Education, Katowice, Poland
Locations (1):
- The Jerzy Kukuczka Academy of Physical Education, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD.

REFERENCES:
- [Derived] Filip-Stachnik A, Krzysztofik M, Del Coso J, Palka T, Sadowska-Krepa E. The Effect of Acute Caffeine Intake on Resistance Training Volume, Prooxidant-Antioxidant Balance and Muscle Damage Markers Following a Session of Full-Body Resistance Exercise in Resistance-Trained Men Habituated to Caffeine. J Sports Sci Med. 2023 Sep 1;22(3):436-446. doi: 10.52082/jssm.2023.436. eCollection 2023 Sep. PMID 37711718